CLINICAL TRIAL: NCT01634217
Title: Dose Escalation Study With Extension of Inducible Regulatory T Cells (iTregs) in Adult Patients Undergoing Non-Myeloablative HLA Identical Sibling Donor Peripheral Blood Stem Cell Transplantation
Brief Title: Inducible Regulatory T Cells (iTregs) in Non-Myeloablative Sibling Donor Peripheral Blood Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012LS019; MT2012-06R (Other: University of Minnesota Bone Marrow Transplant Program)
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Non-Hodgkin Lymphoma; Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Multiple Myeloma; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Administered 3 x 10^6 iTregs/kg infusion
  Interventions: Biological: iTreg
- Cohort 2 (Experimental): Administered 3 x 10^7 iTregs/kg infusion
  Interventions: Biological: iTreg
- Cohort 3 (Experimental): Administered 3 x 10^8 iTregs/kg infusion
  Interventions: Biological: iTreg
- Cohort 4 (Experimental): Administered 10 x 10^8 iTregs/kg infusion
  Interventions: Biological: iTreg
- Cohort 5 Extension (Experimental): Administered 10 x 10^8 iTregs/kg or best available dose using sirolimus/MMF as graft-versus-host disease (GVHD) prophylaxis. Immunosuppression will consist of a combination of sirolimus and mycophenolate mofetil (MMF). Sirolimus will be administered starting at day -3 with 8mg-12mg oral loading dose followed by single dose 4 mg/day. MMF will be administered starting on day -3 at a dose of 3 gram/day divided in 2 or 3 doses. Intravenous (IV) route between days -3 and +5, then may change to PO between days +6 and +30. Stop MMF at day +30 or 7 days after engraftment, whichever day is later, if no acute GVHD.
  Interventions: Biological: iTreg

INTERVENTIONS:
Biological: iTreg — The iTregs will be infused at the assigned dose without a filter or pump slowly by gravity over 15-60 minutes. The iTregs should be given at least 4 hours before the peripheral blood stem cell (PBSC) infusion (MT2001-10).

SUMMARY:
This is a phase I single center dose escalation study with an extension at the best available dose to determine the tolerability of inducible regulatory T cells (iTregs) when given to adult patients undergoing non-myeloablative HLA-identical sibling donor peripheral blood stem cell (PBSC) transplantation for the treatment of a high risk malignancy. Up to 5 dose cohorts will be tested. Once the tolerable dose is determined for iTregs, enrollment will continue with an additional 10 patients using sirolimus/Mycophenolate mofetil (MMF) graft-versus-host disease (GVHD) prophylaxis to gain further safety information and to provide pilot data in this treatment setting.

DETAILED DESCRIPTION:
Co-enrollment in University Of Minnesota protocol MT2001-10 is required and transplantation will be according to that protocol with iTregs administered the morning of day 0 followed no sooner than 4 hours later by the PBSC transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years of age with an HLA-identical sibling donor
* One of the following disease categories:

  * Acute myelogenous leukemia - high risk CR1 (as evidenced by preceding MDS, intermediate to high risk cytogenetics, ≥ 2 cycles to obtain CR, erythroblastic or megakaryocytic leukemia; CR2+. All patients must be in CR as defined by hematological recovery (ANC > 0.5x 109/L), AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
  * Acute lymphocytic leukemia - high risk CR1 [t(9;22), t (1:19), t(4;11) or other MLL rearrangements] or >1cycle to obtain CR; CR2+. All patients must be in CR as defined by hematological recovery (ANC > 0.5x 109/L), AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
  * Chronic myelogenous leukemia all types except blast crisis (note treated blast crisis in chronic phase is eligible)
  * Non-Hodgkin lymphoma or Hodgkin lymphoma demonstrating chemosensitive disease
  * Myelodysplastic syndrome with severe pancytopenia, leading to either transfusion dependency or increased risk for infections
* Performance status: Karnofsky ≥ 60%
* Adequate organ function within 28 days of study enrollment defined as:

  * Liver: SGOT and SGPT < 5.0 x ULN; total bilirubin < 3 x ULN
  * Renal: serum creatinine < 2.0 mg/dl or glomerular filtration rate (GFR) > 40 mL/min/1.73m2. Patients with a creatinine > 1.2 mg/dl or a history of renal dysfunction must have glomerular filtration rate (GFR) > 40 mL/min/1.73m2
  * Albumin: > 2.5 g/dL
  * Cardiac: No decompensated CHF or uncontrolled arrhythmia; ejection fraction > 35% within 6 weeks prior to study enrollment
  * Pulmonary: No O2 requirements; DLCO > 30% predicted within 6 weeks prior to study enrollment
* If recent mold infection (e.g. aspergillus) must have minimum of 30 days of therapy and responsive disease and be cleared by Infectious Disease
* Sexually active females of child bearing potential and males must agree to use effective contraception for the duration of the transplant period
* Voluntary written consent

Exclusion Criteria:

* Pregnancy or breast feeding - women of childbearing potential must have a negative pregnancy test within 28 days of study enrollment.
* Prior myeloablative transplant within previous 3 months of study enrollment.
* Evidence of HIV infection or known HIV positive serology.
* Active serious infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3-5 infusional toxicity | Within 48 Hours After iTregs Administration
  Targeted adverse events and unexpected events not explained by the PBSCT or disease will be collected [(1-4 hours after the iTreg infusion and before the PBSCT at day 0) and 24 hours and 48 hours after the iTreg infusion (+/- 2 hours)]

SECONDARY OUTCOMES:
Cumulative incidence of grade II-IV acute graft-versus-host disease (GVHD) | Day 100
  Graft-versus-host disease (GVHD) is a complication that can occur after a stem cell or bone marrow transplant in which the newly transplanted material attacks the transplant recipient's body. Abstracted from the routine clinical data collected for the primary transplant protocol (MT2001-10).
Incidence of chronic graft-versus-host disease (GVHD) | 12 Months
  Graft-versus-host disease (GVHD) is a complication that can occur after a stem cell or bone marrow transplant in which the newly transplanted material attacks the transplant recipient's body. Abstracted from the routine clinical data collected for the primary transplant protocol (MT2001-10).
Relapse of Disease | 12 Months
  The return of signs and symptoms of a disease after a remission.
Survival | 1 Year
  Number (count) of patients alive at 1 year after treatment.
Survival | Day 100
  Number (count) of patients alive at Day 100.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] MacMillan ML, Hippen KL, McKenna DH, Kadidlo D, Sumstad D, DeFor TE, Brunstein CG, Holtan SG, Miller JS, Warlick ED, Weisdorf DJ, Wagner JE, Blazar BR. First-in-human phase 1 trial of induced regulatory T cells for graft-versus-host disease prophylaxis in HLA-matched siblings. Blood Adv. 2021 Mar 9;5(5):1425-1436. doi: 10.1182/bloodadvances.2020003219. PMID 33666654